CLINICAL TRIAL: NCT00448266
Title: Randomized Phase II/III Study of Intensified Alkylating Agent Chemotherapy With Peripheral Blood Progenitor Cell Support in the Preoperative Chemotherapy of Breast Tumors That Are Deficient for Homologous Recombination.
Brief Title: Intensified IAA With PBPC Support in Breast Tumors With Evidence of a HRD
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Activation of a similar multicenter study for same population
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Prof. Dr. S. Rodenhuis, NKI-AVL
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N06IAA
Record Dates: First submitted 2007-03-14; First posted 2007-03-16 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2010-10

CONDITIONS: Breast Cancer
Keywords: Breast cancer; high-dose chemotherapy; Homologous Recombination Deficiency; Alkylator therapy; Peripheral Blood Progenitor Cell Support
MeSH Terms: conditions — Breast Neoplasms | interventions — Carboplatin; Thiotepa; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Experimental): 1 course ddAc, 2 courses IAA with PBPC support
  Interventions: Drug: Intensified Cyclophophamide, Carboplatin and Thiotepa
- 1 (Active Comparator): 3 courses ddAC
  Interventions: Drug: dose dense adriamycine and cyclophosphamide

INTERVENTIONS:
Drug: Intensified Cyclophophamide, Carboplatin and Thiotepa — 2 courses of Intensified Cyclophophamide, Carboplatin and Thiotepa with PBPC support
  Arms: 2
Drug: dose dense adriamycine and cyclophosphamide — dose dense adriamycine and cyclophosphamide, Q 2 weeks
  Arms: 1

SUMMARY:
This phase II/III trial will investigate the ability of chemotherapy with 'Intensified Aklylating Agents (IAA) to achieve a high pathological complete response (pCR) rate when employed in the preoperative chemotherapy of breast cancer with evidence of a Homologous Recomination Deficiency (HRD).

DETAILED DESCRIPTION:
This phase II/III trial will investigate the ability of chemotherapy with 'Intensified Alkylating Agents' (IAA) to achieve a high pathological complete response (pCR) rate when employed in the preoperative chemotherapy of breast cancer with evidence of a Homologous Recombination Deficiency (HRD).

Homologous Recombination (HR) is a DNA repair mechanism that can repair double-strand DNA breaks. It is the only reliable repair mechanism that can repair the consequences of DNA adducts caused by bifunctional alkylating agensts (such as cyclophosphamide, thiotepa or carboplatin). Alternative DNA repair mechanisms are available in case of HRD, but these induce DNA mutations and chromosome aberrations and thus give rise to major genetic instability. HRD is a consequence of inactivation of BRCA-1 or BRCA-2, but may also be caused by defects in the Fanconi anemia pathway or by amplification of the EMSY gene. HRD is present in breast cancer cells but not in healthy cells of BRCA-1 or BRCA-2 mutation carriers, and also in up to 30% of sporadic breast cancers.

Patients under 60 years of age with intermediate or high risk breast cancer, whose tumors show evidence of HRD and do not contain a HER2/neu amplification are eligible. All patients will receive 3 courses of standard preoperative chemotherapy with dose-dense Doxorubicin and Cyclophosphamide (ddAC). Patients with a favorable response according to repeat MRI, will be randomized to undergo either a further 3 courses of ddAC prior to local therapy and endocrine adjuvant therapy (standard arm) or 1 course of ddAC followed by peripheral blood progenitor cell (PBPC) harvest and 2 courses of IAA with Cyclophosphamide (3 g/m2), thiotepa (240 mg/m2) and carboplatin (800 mg/m2) (experimental arm). IAA is administered during a 1 or 2-night hospital stay, the bone marrow aplasia phase is managed on an out-patient basis and the second course will be started on day 22 of the first one. Patients who do not achieve a favorable response as determined by their MRI after 3 cycles of ddAC will be offered treatment according to the experimental arm as salvage therapy.

The primary endpoint of the study is the pCR rate of the breast. The phase II part of the study will serve to further develop the pathology tests for HRD and to estimate the pCR rates of HRD-breast cancers to both the conventional and the experimental treatments. The phase III part of the study will be initiated when the test for HRD is sufficiently standardized to be employed in a multi-center setting and when the preliminary information collected at that point continues to be consistent with the assumption that HRD renders tumor cells highly sensitive to IAA. If breast cancer is indeed exquisitely sensitive to IAA, the pCR rate in the experimental arm could rise from 10% to 30% in luminal tumor types and from 50% to 80% in basal-like tumor types. For 80% power to detect such a response-improvement, 186 patients with HRD must be included in the phase III part of the study.

ELIGIBILITY:
* Proven infiltrating breast cancer with either a primary tumor over 3 cm in size (clinical examination) or cytologically proven spread to the axillary lymph nodes.
* Stage II or stage III disease (revised AJCC staging system 2001). Patients with 'locally advanced breast cancer' are consequently eligible, including those with ipsilateral supraclavicular lymph node metastases. In stage II patients with T1N1 disease, N1 status must have been demonstrated by either fine needle aspiration from an axillary lymph node or by a metastasis of over 2 mm in diameter in a sentinel node biopsy. Stage IIA patients without lymph node metastases are only eligible if the tumor is over 3 cms in diameter.
* High-risk disease, according to Adjuvant Online version 8.0: the expected 10-year recurrence-free survival without systemic adjuvant therapy according to this program must be 60% or lower.
* The tumor must be HER2/neu-negative (either score 0 or 1 at immunohistochemistry or negative at in situ hybridization [CISH or FISH] in case of score 2 or 3 at immunohistochemistry).
* The tumor must test positive for homologous recombination deficiency, as defined by the test of the pathology department of the NKI-AVL (M.J. van de Vijver).
* Age 18 to 59 years; patients older than 59 years may be included when considered 'biologically 59 years or younger'.
* Performance status: WHO 0 or I.
* No previous radiation therapy or chemotherapy.
* No other malignancy except carcinoma in situ, unless the other malignancy was treated 5 or more years ago with curative intent without the use of chemotherapy or radiation therapy.
* Adequate bone marrow function (W.B.C. count > 3.0 x 109/l, platelets > 100 x 109/l).
* Adequate hepatic function (ALAT, ASAT and bilirubin < 2 x upper limit of normal).
* Adequate renal function (creatinine clearance > 60 ml/min).
* Radionuclide ejection fraction > 0.50.
* Pregnancy or breast feeding must be excluded and patients must use adequate contraceptive protection.
* No evidence of distant metastases. Staging examinations must have included a chest roentgenogram, an ultrasound examination of the liver and an isotope bone scan. Abnormal uptake on the isotope bone scan can only be accepted if bone metastases were excluded by MRI.
* At randomization, hormone receptor status and HER2/neu receptor status must be known. In case of 2+ HER2/neu expression by immunohistochemistry, FISH or CISH examination is required.
* Informed consent.

Ages: 18 Years to 59 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2007-05; Primary Completion 2010-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Percentage of tumors with HRD (phase II part)
pCR rate

SECONDARY OUTCOMES:
Comparison of extramedullary toxicity between the treatment arms.
Need for hospitalization.
Recurrence-free survival and overall survival (phase III part).

CONTACTS AND LOCATIONS:
Overall Officials: Sjoerd Rodenhuis, Principal Investigator — The Netherlands Cancer Institute
Locations (1):
- NKI-AVL, Amsterdam, Netherlands